CLINICAL TRIAL: NCT03332225
Title: A Personalized Randomized Trial of Validation and Restoration of Immune Dysfunction in Severe Infections and Sepsis
Brief Title: A Trial of Validation and Restoration of Immune Dysfunction in Severe Infections and Sepsis
Acronym: PROVIDE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hellenic Institute for the Study of Sepsis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PROVIDE; 2017-002171-26 (EudraCT Number)
Record Dates: First submitted 2017-10-27; First posted 2017-11-06 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Sepsis; Macrophage Activation Syndrome
Keywords: sepsis; macrophage activation syndrome; immunoparalysis; anakinra; recombinant human interferon-gamma; HLA-DR
MeSH Terms: conditions — Sepsis; Macrophage Activation Syndrome | interventions — Interleukin 1 Receptor Antagonist Protein; Saline Solution

STUDY DESIGN:
Intervention Model Description: Treatment with recombinant human interferon-gamma or anakinra
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anakinra (Experimental): Treatment with iv anakinra 200 mg three times daily (every eight hours) for seven days and sc 1ml N/S 0.9% every other day for 15 days
  Interventions: Drug: Anakinra
- IV Placebo (Placebo Comparator): Treatment with iv 1ml N/S 0.9% three times daily (every eight hours) for seven days and sc 1ml N/S 0.9% every other day for 15 days
  Interventions: Drug: Placebo
- Recombinant human interferon-gamma (Experimental): Treatment with sc recombinant human interferon-gamma every other day for a total of 15 days and with iv 1ml N/S 0.9% three times daily (every eight hours) for seven days
  Interventions: Drug: Recombinant human interferon-gamma

INTERVENTIONS:
Drug: Anakinra — Treatment with anakinra
  Other Names: Kineret
  Arms: Anakinra
Drug: Recombinant human interferon-gamma — Treatment with recombinant human interferon-gamma
  Other Names: Imukin
  Arms: Recombinant human interferon-gamma
Drug: Placebo — Treatment with Placebo
  Other Names: Saline Solution
  Arms: IV Placebo

SUMMARY:
The aim of the study is to conduct one RCT of personalized immunotherapy in sepsis targeting patients who lie either on the predominantly hyper-inflammatory arm or on the predominantly hypo-inflammatory arm of the spectrum of the host response. These patients will be selected by the use of a panel of biomarkers and laboratory findings and they will be randomly allocated to placebo or immunotherapy treatment according to their needs.

DETAILED DESCRIPTION:
Sepsis is a life-threatening organ dysfunction that results from the dysregulated host response to an infection. Accumulating knowledge suggests that this dysregulated host response has a broad spectrum where some patients lie to the two extremes of this spectrum whereas the majority of patients lie in between. The first extreme encompasses patients who are dominated from a hyper-inflammatory response to an infectious insult. On the other extreme lie patients who do not have any hyper-inflammatory response; instead these patients are dominated by an exhausted immune response to an infectious stimulus. The remaining patients have features of both hyper- and hypo-inflammatory responses.

Randomized clinical trials (RCTs) that have investigated the effects of immunotherapy in sepsis have all failed to establish beneficial effects for the patients. The reasons for that are multiple but one of the most important is the current notion that sepsis is a complex disorder with heterogeneity regarding patient characteristics. Thus, it is necessary to try and find ways to personalise the immunomodulatory treatment of sepsis. In the clinical trial proposed here, two personalised approaches will be investigated.

Some 25 years ago, there were high expectations of the blockade of interleukin (IL)-1 in sepsis using the human recombinant IL-1 receptor antagonist, anakinra. The expectations were based on animal experiments as well as positive results in a single-centre clinical trial. However, in a large international trial, anakinra did not show benefit over placebo. Still, it became clear from this study, enrolling 906 patients that intravenous anakinra was a very safe drug: there was neither excess mortality in these critically ill patients, nor increased susceptibility to secondary infections. In a post-hoc analysis of this trial published in 2016, it was demonstrated that a subgroup of 34 patients showed a clinical picture compatible with macrophage activation syndrome. Since bone marrow was not performed in these patients, the investigators prefer to call this macrophage activation like syndrome (MALS). MALS is a dreaded complication with a mortality rate in the order of 70%. The post-hoc analysis showed that patients receiving anakinra had 30% significant survival benefit compared to those receiving placebo. From these data it can be concluded that it is important to recognize patients with this complication of sepsis and that anakinra might be a beneficial drug.

A survey of the database of sepsis patients in the Hellenic Sepsis Study Group revealed that 5% of the patients with septic shock suffered from MALS. It was found in this study that MAS can be easily and reliably diagnosed by measuring ferritin in the blood. A cut off of 4.420ng/ml had specificity more than 97%.

Another important clinical phenomenon in sepsis is that patients may run into a phase of immunoparalysis. In this situation, the immune cells do not produce any more proinflammatory cytokines and switch to production of anti-inflammatory cytokines such as IL-10; they also loose important functional markers such HLA-DR. Patients with immunoparalysis have a 50% risk of dying in the subsequent 28 days. There is evidence from preclinical studies and from the endotoxin challenge model in human volunteers that immunoparalysis is reversible at least to some extent. The best candidate drug for this would be interferon gamma (IFNγ). Immunosuppression established in healthy volunteers after experimental endotoxemia was reversed after administration of recombinant human interferon-gamma (rhIFNγ). rhIFNγ was also investigated for this purpose in nine patients at septic shock in a small open-label and non-randomized clinical trial; reversal of immunoparalysis was achieved. The extensive experience with IFNγ teaches that it is a safe drug, the main side effect being fever and flu-like syndrome, which can be mitigated by premedication with a prostaglandin inhibitor like paracetamol. In patients with autoimmune diseases like systemic lupus erythematosus (SLE) and multiple sclerosis flares of the disease induced by IFNγ have been described. So these diseases are contraindications for the drug.

The purpose of this study is to investigate in a randomised placebo-controlled clinical trial with a double-dummy design in patients with septic shock, whether personalised immunotherapy directed against either MALS or immunoparalysis is able to change the perspective for these critically ill patients.

MALS is considered as a more direct life-threatening manifestation of sepsis than immunoparalysis. For that reason all patients will be randomised with evidence of MALS for anakinra or placebo, irrespective the state of immunity as measured by HLA-DR positivity.

The aim of the study is to conduct one RCT of personalized immunotherapy in sepsis targeting patients who lie either on the predominantly hyper-inflammatory arm or on the predominantly hypo-inflammatory arm of the spectrum of the host response. These patients will be selected by the use of a panel of biomarkers and laboratory findings and they will be allocated to placebo or immunotherapy treatment according to their needs.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or above 18 years
* Male or female gender
* In case of women, unwillingness to remain pregnant during the study period
* Written informed consent provided by the patient or by one first-degree relative/spouse in case of patients unable to consent
* Community-acquired pneumonia or hospital-acquired pneumonia or ventilator-associated pneumonia or primary bacteremia or acute cholangitis
* Sepsis defined by the Sepsis-3 definitions.
* Patients with laboratory diagnosis of MALS or hypo-inflammation (immune-paralysis) based on two consecutive blood sampling with 24 hours apart. MALS is defined as the presence of ferritin >4,420 ng/ml and hypo-inflammation as HLA-DR expression on CD14-monocytes (co-expression) less than 30%

Exclusion Criteria:

* Age below 18 years
* Denial for written informed consent
* Acute pyelonephritis or intraabdominal infection other than AC, meningitis or skin infection. It is explicitly stated that in the case of a patient with both AC and any other type of intraabdominal infection, the patient cannot be enrolled.
* Any stage IV malignancy
* Any do not resuscitate decision
* In the case of BSI, patients with blood cultures growing coagulase-negative staphylococci or skin commensals or catheter-related infections cannot be enrolled.
* Active tuberculosis (TB) as defined by the co-administration of drugs for the treatment of TB
* Infection by the human immunodeficiency virus (HIV)
* Any primary immunodeficiency
* Oral or IV intake of corticosteroids at a daily dose equal or greater than 0.4 mg prednisone or greater the last 15 days
* Any anti-cytokine biological treatment the last one month
* Medical history of systemic lupus erythematosus
* Medical history of multiple sclerosis or any other demyelinating disorder
* Pregnancy or lactation. Women of child-bearing potential will be screened by a urine pregnancy test before inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality | 28 days
  Mortality will be compared between the groups of treatment

SECONDARY OUTCOMES:
Mortality | 90 days
  Mortality will be compared between the groups of treatment
Time to decrease of SOFA score by more than 50% | 28 days
  The time to decrease of SOFA score by more than 50% will be compared between the groups of treatment
Time to infection resolution | 28 days
  The time to infection resolution will be compared between the groups of treatment
Duration of hospitalisation | 28 days
  The duration of hospitalisation will be compared between the groups of treatment
Number of secondary infections | 28 days
  The number of secondary infections will be compared between the groups of treatment
Cytokine stimulation | 4 days
  Cytokine stimulation from peripheral blood mononuclear cells will be compared between the groups of treatment
Cytokine stimulation | 7 days
  Cytokine stimulation from peripheral blood mononuclear cells will be compared between the groups of treatment
Gene expression | 7 days
  Gene expression of peripheral blood mononuclear cells will be compared between the groups of treatment
Gut microbiome changes | 7 days
  Gut microbiome changes will be compared between the groups of treatment
Epigenetic changes | 7 days
  Epigenetic changes of circulating monocytes will be compared between the groups of treatment
Classification of the immune function | 28 days
  Classification of the immune function of screened patients not characterized with MALS neither with hypo-inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Antonios Papadopoulos, MD, PhD, Principal Investigator — National Kapodistrian University of Athens, Medical School
Locations (13):
- Greece (13):
  - 2nd Department of Critical Care Medicine, Athens, Haidari
  - 4th Department of Internal Medicine, Athens, Haidari
  - Intensive Care Unit, Ioannina University Hospital, Ioannina, Ioannina
  - Intensive Care Unit, Center for Accident Rehabilitation (KAT) of Athens, Athens, Kifissia
  - Department of Internal Medicine, Patras University Hospital, Pátrai, Rion
  - Intensive Care Unit, Alexandroupolis University Hospital, Alexandroupoli
  - 1st Department of Pulmonary Medicine and Intensive Care Unit, Athens
  - Intensive Care Unit, "Latsio", Thriasio Elefsis General Hospital, Elefsina
  - Intensive Care Unit, "Koutlimbaneio & Triantafylleio" Larissa General Hospital, Larissa
  - Department of Internal Medicine, Larissa University Hospital, Larissa
  - Intensive Care Unit, "Tzanio" Piraeus General Hospital, Piraeus
  - Intensive Care Unit, "Aghios Dimitrios" Thessaloniki General Hospital, Thessaloniki
  - Intensive Care Unit, "G.Gennimatas" Thessaloniki General Hospital, Thessaloniki

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Result] Opal SM, Fisher CJ Jr, Dhainaut JF, Vincent JL, Brase R, Lowry SF, Sadoff JC, Slotman GJ, Levy H, Balk RA, Shelly MP, Pribble JP, LaBrecque JF, Lookabaugh J, Donovan H, Dubin H, Baughman R, Norman J, DeMaria E, Matzel K, Abraham E, Seneff M. Confirmatory interleukin-1 receptor antagonist trial in severe sepsis: a phase III, randomized, double-blind, placebo-controlled, multicenter trial. The Interleukin-1 Receptor Antagonist Sepsis Investigator Group. Crit Care Med. 1997 Jul;25(7):1115-24. doi: 10.1097/00003246-199707000-00010. PMID 9233735
- [Result] Shakoory B, Carcillo JA, Chatham WW, Amdur RL, Zhao H, Dinarello CA, Cron RQ, Opal SM. Interleukin-1 Receptor Blockade Is Associated With Reduced Mortality in Sepsis Patients With Features of Macrophage Activation Syndrome: Reanalysis of a Prior Phase III Trial. Crit Care Med. 2016 Feb;44(2):275-81. doi: 10.1097/CCM.0000000000001402. PMID 26584195
- [Result] Kyriazopoulou E, Leventogiannis K, Norrby-Teglund A, Dimopoulos G, Pantazi A, Orfanos SE, Rovina N, Tsangaris I, Gkavogianni T, Botsa E, Chassiou E, Kotanidou A, Kontouli C, Chaloulis P, Velissaris D, Savva A, Cullberg JS, Akinosoglou K, Gogos C, Armaganidis A, Giamarellos-Bourboulis EJ; Hellenic Sepsis Study Group. Macrophage activation-like syndrome: an immunological entity associated with rapid progression to death in sepsis. BMC Med. 2017 Sep 18;15(1):172. doi: 10.1186/s12916-017-0930-5. PMID 28918754
- [Result] Leentjens J, Kox M, Koch RM, Preijers F, Joosten LA, van der Hoeven JG, Netea MG, Pickkers P. Reversal of immunoparalysis in humans in vivo: a double-blind, placebo-controlled, randomized pilot study. Am J Respir Crit Care Med. 2012 Nov 1;186(9):838-45. doi: 10.1164/rccm.201204-0645OC. Epub 2012 Jul 19. PMID 22822024
- [Result] Docke WD, Randow F, Syrbe U, Krausch D, Asadullah K, Reinke P, Volk HD, Kox W. Monocyte deactivation in septic patients: restoration by IFN-gamma treatment. Nat Med. 1997 Jun;3(6):678-81. doi: 10.1038/nm0697-678. PMID 9176497
- [Result] Calandra T, Cohen J; International Sepsis Forum Definition of Infection in the ICU Consensus Conference. The international sepsis forum consensus conference on definitions of infection in the intensive care unit. Crit Care Med. 2005 Jul;33(7):1538-48. doi: 10.1097/01.ccm.0000168253.91200.83. PMID 16003060
- [Result] Christ-Crain M, Jaccard-Stolz D, Bingisser R, Gencay MM, Huber PR, Tamm M, Muller B. Effect of procalcitonin-guided treatment on antibiotic use and outcome in lower respiratory tract infections: cluster-randomised, single-blinded intervention trial. Lancet. 2004 Feb 21;363(9409):600-7. doi: 10.1016/S0140-6736(04)15591-8. PMID 14987884
- [Result] Kalil AC, Metersky ML, Klompas M, Muscedere J, Sweeney DA, Palmer LB, Napolitano LM, O'Grady NP, Bartlett JG, Carratala J, El Solh AA, Ewig S, Fey PD, File TM Jr, Restrepo MI, Roberts JA, Waterer GW, Cruse P, Knight SL, Brozek JL. Management of Adults With Hospital-acquired and Ventilator-associated Pneumonia: 2016 Clinical Practice Guidelines by the Infectious Diseases Society of America and the American Thoracic Society. Clin Infect Dis. 2016 Sep 1;63(5):e61-e111. doi: 10.1093/cid/ciw353. Epub 2016 Jul 14. PMID 27418577
- [Result] Zilberberg MD, Shorr AF. Ventilator-associated pneumonia: the clinical pulmonary infection score as a surrogate for diagnostics and outcome. Clin Infect Dis. 2010 Aug 1;51 Suppl 1:S131-5. doi: 10.1086/653062. PMID 20597663
- [Result] Giamarellos-Bourboulis EJ, Tsaganos T, Tsangaris I, Lada M, Routsi C, Sinapidis D, Koupetori M, Bristianou M, Adamis G, Mandragos K, Dalekos GN, Kritselis I, Giannikopoulos G, Koutelidakis I, Pavlaki M, Antoniadou E, Vlachogiannis G, Koulouras V, Prekates A, Dimopoulos G, Koutsoukou A, Pnevmatikos I, Ioakeimidou A, Kotanidou A, Orfanos SE, Armaganidis A, Gogos C; Hellenic Sepsis Study Group. Validation of the new Sepsis-3 definitions: proposal for improvement in early risk identification. Clin Microbiol Infect. 2017 Feb;23(2):104-109. doi: 10.1016/j.cmi.2016.11.003. Epub 2016 Nov 14. PMID 27856268
- [Result] Pontikis K, Karaiskos I, Bastani S, Dimopoulos G, Kalogirou M, Katsiari M, Oikonomou A, Poulakou G, Roilides E, Giamarellou H. Outcomes of critically ill intensive care unit patients treated with fosfomycin for infections due to pandrug-resistant and extensively drug-resistant carbapenemase-producing Gram-negative bacteria. Int J Antimicrob Agents. 2014 Jan;43(1):52-9. doi: 10.1016/j.ijantimicag.2013.09.010. Epub 2013 Oct 16. PMID 24183799
- [Derived] Kranidioti E, Ricano-Ponce I, Antonakos N, Kyriazopoulou E, Kotsaki A, Tsangaris I, Markopoulou D, Rovina N, Antoniadou E, Koutsodimitropoulos I, Dalekos GN, Vlachogianni G, Akinosoglou K, Koulouras V, Komnos A, Kontopoulou T, Dimopoulos G, Netea MG, Kumar V, Giamarellos-Bourboulis EJ. Modulation of Metabolomic Profile in Sepsis According to the State of Immune Activation. Crit Care Med. 2024 Nov 1;52(11):e536-e544. doi: 10.1097/CCM.0000000000006391. Epub 2024 Aug 23. PMID 39418210
- [Derived] Leventogiannis K, Kyriazopoulou E, Antonakos N, Kotsaki A, Tsangaris I, Markopoulou D, Grondman I, Rovina N, Theodorou V, Antoniadou E, Koutsodimitropoulos I, Dalekos G, Vlachogianni G, Akinosoglou K, Koulouras V, Komnos A, Kontopoulou T, Prekates A, Koutsoukou A, van der Meer JWM, Dimopoulos G, Kyprianou M, Netea MG, Giamarellos-Bourboulis EJ. Toward personalized immunotherapy in sepsis: The PROVIDE randomized clinical trial. Cell Rep Med. 2022 Nov 15;3(11):100817. doi: 10.1016/j.xcrm.2022.100817. PMID 36384100
- [Derived] Karakike E, Giamarellos-Bourboulis EJ. Macrophage Activation-Like Syndrome: A Distinct Entity Leading to Early Death in Sepsis. Front Immunol. 2019 Jan 31;10:55. doi: 10.3389/fimmu.2019.00055. eCollection 2019. PMID 30766533